CLINICAL TRIAL: NCT07233733
Title: Efficacy of Connective Tissue Graft Wall Technique and Enamel Matrix Derivative in the Regenerative Treatment of Intrabony Periodontal Defects: A Prospective Clinical Study
Brief Title: A Clinical Study of Connective Tissue Graft and Enamel Matrix Derivative in the Treatment of Intrabony Periodontal Defects
Acronym: CTG + EMD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Phạm Đình Thiên Khải (Other)
Collaborators: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Sponsor-Investigator, Phạm Đình Thiên Khải, Resident Doctor in Periodontology, Principal Investigator, University of Medicine and Pharmacy at Ho Chi Minh City
Organization: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: No. 716/HĐĐĐ-ĐHYD; 258/2025/HĐ-ĐHYD (Other Grant/Funding Number: University of Medicine and Pharmacy at Ho Chi Minh City)
Record Dates: First submitted 2025-09-26; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Periodontal Diseases; Regeneration
Keywords: connective tissue; Enamel Matrix Derivative (EMD); Periodontal Regeneration; Infrabony Defects
MeSH Terms: conditions — Periodontal Diseases | interventions — Debridement; Edetic Acid; emerin; Suture Techniques; Amoxicillin; Clavulanic Acid; Ibuprofen

STUDY DESIGN:
Intervention Model Description: This is a single-arm interventional clinical trial in which all enrolled patients receive periodontal regenerative surgery using the connective tissue graft wall technique combined with enamel matrix derivative (Emdogain®). The model was selected to evaluate clinical and radiographic outcomes of this specific surgical approach without a comparator group
Masking Description: Outcome assessors were blinded to the surgical intervention. Examiners responsible for clinical and radiographic measurements were not involved in the surgical procedures and were unaware of the treatment allocation, ensuring unbiased data collection
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Connective Tissue Wall + Enamel Matrix Derivative (Experimental): Periodontal regenerative surgery using a connective tissue graft (CTG) "soft-tissue wall" combined with enamel matrix derivative (EMD, Emdogain®) under a minimally invasive flap design.
  Interventions: Procedure: Connective Tissue Graft (CTG) Wall Technique; Procedure: Minimally Invasive Flap Design; Procedure: Root Surface Preparation and Debridement; Biological: Growth Factor Application (EDTA + EMD); Procedure: Suturing Technique; Drug: Amoxicillin/Clavulanate Potassium 875 MG-125 MG Oral Tablet; Drug: Ibuprofen (Advil); Drug: chlorhexidine mouthrinse

INTERVENTIONS:
Procedure: Connective Tissue Graft (CTG) Wall Technique — After flap elevation and thorough degranulation/root debridement, a palatal connective tissue graft is harvested with the four-incision technique, de-epithelialized, and adapted to the buccal flap to create a stable soft-tissue wall.
  Other Names: Connective Tissue Graft Wall Technique
Procedure: Minimally Invasive Flap Design — Split-thickness vestibular releasing flap with external papilla reflection to allow coronal advancement and preserve blood supply.
Procedure: Root Surface Preparation and Debridement — Thorough degranulation and root surface debridement using ultrasonic and hand instruments; intraoperative recording of defect depth and morphology.
Biological: Growth Factor Application (EDTA + EMD) — Conditioning of the root surface with 24% EDTA gel for 2 minutes, rinsing, followed by application of enamel matrix derivative (EMD; Emdogain®) to the root surface and into the intrabony defect.
Procedure: Suturing Technique — Combination of horizontal mattress and interrupted sutures to achieve tension-free primary closure.
Drug: Amoxicillin/Clavulanate Potassium 875 MG-125 MG Oral Tablet — 875/125 mg orally, twice daily for 5 days, prescribed as postoperative antibiotic therapy.
Drug: Ibuprofen (Advil) — 400 mg orally, three times daily for 5 days, prescribed for postoperative pain and inflammation control.
Drug: chlorhexidine mouthrinse — 0.12% solution, twice daily for 2 weeks, prescribed for chemical plaque control.

SUMMARY:
This clinical study aims to evaluate the effectiveness of periodontal regenerative surgery using the connective tissue graft (CTG) wall technique combined with enamel matrix derivative (EMD) in patients who have intrabony periodontal defects. The purpose is to determine whether this combined approach can enhance both bone regeneration and soft-tissue stability compared with the patient's initial condition.

Eligible participants will receive periodontal surgery in which a connective tissue graft and enamel matrix derivative are applied to the defect site. The study will monitor clinical improvements such as attachment gain, reduction in pocket depth, bone fill observed on cone-beam computed tomography (CBCT), and stability of the gingival margin and soft-tissue thickness. Clinical parameters (probing depth and attachment level) are recorded at baseline, 3 months, and 6 months. Gingival and hygiene parameters (recession, gingival thickness, plaque, and bleeding scores) are assessed at baseline, 1 month, 3 months, and 6 months. Radiographic bone outcomes are measured at baseline and 6 months, and early wound healing is assessed at 1 and 2 weeks.

The main goal is to assess whether CTG + EMD treatment provides predictable periodontal regeneration, improved tissue stability, and better esthetic outcomes for patients with periodontitis.

DETAILED DESCRIPTION:
This is a prospective, single-group interventional clinical trial conducted at the University of Medicine and Pharmacy at Ho Chi Minh City to evaluate the effectiveness of the connective tissue graft (CTG) wall technique combined with enamel matrix derivative (EMD, Emdogain®, Straumann) in the regenerative treatment of intrabony periodontal defects. The study included 17 patients diagnosed with stage III-IV periodontitis who presented with radiographically confirmed intrabony defects suitable for regenerative therapy.

All participants received treatment following a standardized periodontal surgical protocol. After local anesthesia, a split-thickness vestibular releasing flap was prepared to allow coronal advancement, with external reflection of the papilla at the defect site. Thorough degranulation and root surface debridement were performed using ultrasonic and hand instruments. The root surface was conditioned with 24% EDTA gel for 2 minutes, rinsed with saline, and then enamel matrix derivative was applied onto the root surface and into the defect. A palatal connective tissue graft harvested using the four-incision technique was de-epithelialized, trimmed to span the papillae, and sutured to the buccal flap to form a stable soft-tissue wall. The flap was coronally advanced and secured with horizontal mattress and interrupted sutures to achieve tension-free primary closure.

Clinical and radiographic outcomes are evaluated at multiple time points.

Clinical parameters: probing pocket depth (PPD) and clinical attachment level (CAL) at baseline, 3 months, and 6 months.

Soft-tissue and hygiene parameters: gingival recession (buccal and interproximal), gingival thickness, full-mouth plaque score (FMPS), and full-mouth bleeding score (FMBS) at baseline, 1, 3, and 6 months.

Radiographic parameters: infrabony defect depth, buccal bone dehiscence, suprabony component, and defect angle measured on cone-beam computed tomography (CBCT) at baseline and 6 months.

Early wound healing: assessed at 1 and 2 weeks using the Early Healing Index (EHI).

The study was conducted at the Department of Periodontology, University of Medicine and Pharmacy at Ho Chi Minh City, between June 2024 and August 2025. The protocol was reviewed and approved by the Institutional Review Board of the University of Medicine and Pharmacy at Ho Chi Minh City (Approval No. 716/HĐĐĐ-ĐHYD, dated June 13, 2024). All participants provided written informed consent before enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years old who can provide written informed consent.
* Diagnosis of stage III-IV periodontitis (2017 World Workshop).
* Completed initial non-surgical periodontal therapy with good plaque control.
* Full-mouth plaque score (FMPS) ≤20% and full-mouth bleeding score (FMBS) ≤20%.
* Presence of ≥1 intrabony periodontal defect with an intrabony component ≥3 mm, confirmed clinically and radiographically.
* Probing pocket depth (PPD) at the study site ≥6 mm.

Exclusion Criteria:

* Systemic conditions or medications that could affect periodontal healing (e.g., diabetes mellitus, immunodeficiency, bisphosphonates, corticosteroids, immunosuppressants).
* Current smokers or former heavy smokers.
* Pregnancy or lactation.
* Teeth with untreated endodontic lesions or non-vital status; furcation involvement class II-III.
* Untreated occlusal trauma or tooth mobility grade II-III.
* Third molars.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Clinical Attachment Level (CAL) Gain | Baseline 3 months, and 6 months post-surgery
  Change in clinical attachment level measured at the treated intrabony periodontal defect, measured with UNC-15 probe and acrylic stent. The CAL is recorded as the distance from the cementoenamel junction (CEJ) to the base of the periodontal pocket. Unit: millimeters (mm). Negative change = gain (better).
Recession Interproximal (RECi) | Baseline, one month, 3 months, 6 months
  Distance from the cusp tip or incisal edge to the interproximal gingival margin, measured in millimeters, to evaluate changes in papillary and proximal soft tissue level after treatment. Unit: millimeters (mm). Higher = worse.
Radiographic Intrabony Defect Fill (mm) | Baseline and 6 months post-surgery
  Change in vertical depth of the intrabony periodontal defect measured on CBCT at the treated site. Linear distance from the alveolar crest to the base of the defect along the root surface is recorded; greater positive values indicate more defect fill. Unit: millimeters (mm). Positive fill = better.
Recession Buccal (RECb) | Baseline, 1 month, 3 months, and 6 months post-surgery
  Distance from the cusp tip or incisal edge to the buccal gingival margin (zenith point), measured in millimeters, to evaluate changes in papillary and proximal soft tissue level after treatment. Unit: millimeters (mm). Higher = worse.
Probing Pocket Depth (PPD) | Baseline, 3 months, and 6 months
  Distance from gingival margin to base of pocket with UNC-15 probe and stent. Negative change = reduction (better).

SECONDARY OUTCOMES:
Gingival Thickness | Baseline, 3 months, 6 months
  Buccal gingival thickness measured mid-facially using probe transparency method as described by Kan et al. (2003). Unit: categorical (thin / thick). Thick = better.
Early Healing Index (EHI) | 1 week, 2 weeks post-surgery
  Early wound healing quality assessed according to Wachtel (2003) index. Unit: ordinal scale (1-5). 1 = best, 5 = worst.
Full-Mouth Plaque Score (FMPS) | Baseline, 1 month, 3 months, 6 months
  Percentage of tooth surfaces with visible plaque after probing, assessed according to O'Leary et al. (1972). Unit: percentage (%). Lower = better.
Full-Mouth Bleeding Score (FMBS) | Baseline, 1 month, 3 months, 6 months
  Percentage of tooth surfaces with bleeding after probing, assessed according to O'Leary et al. (1972). Unit: percentage (%). Lower = better.
Defect Angle | Baseline and 6 months.
  Calculated as the angle formed between the root surface and bone crest at the defect site on CBCT images. Unit: degrees (°). Descriptive.
Buccal Bone Dehiscence | Baseline, 6 months.
  Vertical distance from CEJ to the most apical part of buccal bone crest measured on CBCT to assess buccal bone resorption. Unit: millimeters (mm). Lower = better.
Suprabony Component | Baseline, 6 months
  Distance from CEJ to alveolar bone crest measured on CBCT; indicates vertical bone loss height. Unit: millimeters (mm).
Infrabony Defect Depth | Baseline, 6 months
  Distance from the cemento-enamel junction (CEJ) to the base of the defect measured on CBCT; used to calculate defect depth. Unit: millimeters (mm). Descriptive
Sex/Gender | At baseline
  Male and Female
Age | At baseline
  Adults, 18 years and older. Unit: years
Defect Depth at Surgery | At surgery
  Distance from bonecrest to base of defect measured intraoperatively in mm
Number of Remaining Bony Walls | At surgery and baseline
  Number of residual bony walls at the intrabony defect, assessed intraoperatively. This classification follows the standard defect morphology description used by Tonetti et al. (1993, 1996). A lower number of walls indicates a less favorable prognosis, while a higher number indicates better regenerative potential.
Defect Location | At baseline
  Categorical (Maxilla / Mandible).
Tooth Type | At baseline
  Categorical (Incisor / Canine / Premolar / Molar).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Medicine and Pharmacy at Ho Chi Minh City - Faculty of Odonto-Stomatology, Ho Chi Minh City, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No